CLINICAL TRIAL: NCT07143162
Title: YOGA-FIT: Protocol for a Crossover Trial Investigating the Feasibility and Impact of Virtual Versus In-person Yoga for Late Subacute & Chronic Stroke Survivors
Brief Title: YOGA-FIT: Investigating the Feasibility and Impact of Virtual Versus In-person Yoga for Late Subacute & Chronic Stroke Survivors
Acronym: YOGA-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Adria Quigley, Assistant Professor, Dalhousie University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: YOGA-FIT
Record Dates: First submitted 2025-08-07; First posted 2025-08-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Stroke; Yoga; LoveYourBrain; Virtual rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person LoveYourBrain Yoga (Experimental): Participants will engage in a 90-minute in-person class that will consist of 10 minutes of breathing, 45 minutes of Yoga postures, 15 minutes of meditation, and 20 minutes of psychoeducation and discussion. Additionally, participants will complete a 45- to 60-minute recorded class on their own time.
  Interventions: Behavioral: LoveYourBrain Yoga
- Virtual LoveYourBrain Yoga (Experimental): Participants will engage in a 90-minute virtual class that will consist of 10 minutes of breathing, 45 minutes of Yoga postures, 15 minutes of meditation, and 20 minutes of psychoeducation and discussion. Additionally, participants will complete a 45- to 60-minute recorded class on their own time.
  Interventions: Behavioral: LoveYourBrain Yoga

INTERVENTIONS:
Behavioral: LoveYourBrain Yoga — The LoveYourBrain Yoga program consists of various techniques, including: breathing, Yoga postures, meditation, and psychoeducation as well as a group discussion.

SUMMARY:
The main objective of this mixed-methods pilot crossover study is to determine the feasibility of virtual and in-person LYB Yoga for adult stroke survivors in Nova Scotia who are at least three months post stroke or more.

The secondary objective is to estimate the efficacy of virtual and in-person yoga for improving balance, walking, mobility, mental health (anxiety and depression), and other health outcomes (pain, sleep, health perception, and falls).

The tertiary objective is to estimate the extent to which cognitive function, fatigue, and health-related quality of life co-evolve with our secondary outcomes.

Participants will engage in LYB Yoga virtual and in-person classes for 90 minutes each, twice per week, as well as one 60-minute recorded class completed on their own time.

DETAILED DESCRIPTION:
LoveYourBrain (LYB) is a six-week manualized Yoga program that was originally developed for traumatic brain injury (TBI) patients. The sessions involve meditation, breathing, a variety of Yoga postures, and psychoeducation and discussion components. The program contains key aspects of neuroplasticity and motor learning, which are essential for promoting stroke recovery.

This program can be adapted to suit the needs of the subacute and chronic stroke survivor population: adjusting postures to allow for hemi-paretic stroke survivor participation, as well as a variety of seated and standing options will be made available in the LYB Yoga program. This program will also involve group discussion, educational activities, and coping strategies to help with stroke recovery, while creating a sense of community and mutual understanding.

The program has not yet been offered in the stroke context, nor is it available across Nova Scotia. Therefore, the main aim of this study is to test the feasibility of adapting LYB for the stroke context and making it widely available across Nova Scotia in a virtual and in-person format.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible if they are an adult (aged 18 or older) late subacute or chronic survivor (minimum of three-months post stroke), residing in Nova Scotia, capable of walking 10-metres or more independently or with supervision or the use of an aid or orthotic, and medically stable for eight weeks prior to the baseline visit. Participants must also be able to follow a three-step command.

Exclusion Criteria:

Participants with severe neglect or other issues affecting their safety and participation will be excluded. Participants with cardiovascular, orthopedic, or neurological diseases other than stroke, impacting walking, balance, and mobility will be excluded. Participants who do not have a stable and reliable internet connection will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Baseline
  Percentage of eligible stroke survivors approached and agree to participate.
Participant satisfaction | Weekly satisfaction questionnaire (weeks 1-24) via smartphone app
  Satisfaction questionnaire
Participant and assessor burden | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Assessment time
Adherence | Weeks 1-24
  Class attendance- Weekly surveys via smartphone app and yoga instructor tracking
Equipment | Weeks 1-24 and interviews at the end of 24 weeks
  Technical issues during virtual classes- Yoga instructor tracking during each class and interviews at the end of the study
Smartphone application | Weeks 1-24 and interviews at the end of 24 weeks
  Issues with smartphone application-Weekly smartphone surveys and interviews at the end of the study
Safety -Serious Adverse Events | Monitoring during each class (weeks 1-24) and at all 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Serious adverse events related to the study

SECONDARY OUTCOMES:
Balance | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Dynamic balance will be assessed using the MiniBESTest
Walking | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Walking speed will be assessed using the 10-metre walking test
Mobility | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Functional mobility will be measured using the 5-times sit-to-stand test
Mental health | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Mental health related outcomes will be measured using the Patient Health Questionnaire (PHQ-9). Scores of 0-4 represent no mental health related concerns, while scores of 4-27 indicate mild-severe depression symptoms on the PHQ-9.
Mental health | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Mental health related outcomes will be measured using the Patient Health Questionnaire (PHQ-9) and General Anxiety Disorder-7 scale. Scores of 0-4 represent no mental health related concerns, while scores of 4-27 indicate mild- severe anxiety or depression symptoms in the PHQ-9. Scores of 0-4 indicate no anxiety, while scores of 5-21 indicate mild-severe symptoms of generalized anxiety on the GAD-7 scale.
Health outcomes | Weekly surveys via smartphone app
  The levels of sleep, pain and health perception will be assessed using the Visual Analog Scale, as well as a question about the number of times the person fell within the past week.

OTHER OUTCOMES:
Cognition | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Cognitive function will be assessed using two executive function (n-back and shifting) tests from the Dalhousie Computerized Attention Battery (DalCAB), a digital self-administered cognitive battery.
Health-related quality of life | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Health-related quality of life will be measured using the European Quality of Life Five Dimension (EQ-5D). Participants will rate the 5 items on a 3-point scale with the resulting index score ranging from 0-1 where 0 is the worst health imaginable and 1 is full health. Using the EQ-VAS, participants rate their health on a vertical visual analogue scale labelled from 0-100, with higher scores reflecting better health.
Post-stroke fatigue | During the 4 assessments (Baseline, 6 weeks, 18 weeks, 24 weeks)
  Fatigue severity will be assessed using the Fatigue Severity Scale-7. A 9-item self-reported questionnaire with a maximum score of 63 where higher scores reflect worse fatigue and impact on daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroCommons, Halifax, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be shared upon request.